CLINICAL TRIAL: NCT04944979
Title: A Phase III, Open-label, Prospective, Multicenter Study to Assess Efficacy, Safety, and Pharmacokinetics of Kedrion Intravenous Human Normal Immunoglobulin (IVIg) 10% in Pediatric Patients Affected by Primary Immunodeficiency Disease (PID)
Brief Title: Clinical Assessment of Pharmacokinetics, Efficacy, and Safety of 10% IVIg in Pediatric PID Patients (KIDCARES10)
Acronym: KIDCARES10
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB070
Record Dates: First submitted 2021-06-11; First posted 2021-06-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Primary Immunodeficiency Disease
Keywords: Immunoglobulin; Kedrion IVIG 10%; IgG Antibodies; Agammaglobulinemia; Hypogammaglobulinemia; Pediatric
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Agammaglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Kedrion IVIG 10% (Experimental): Participants will receive intravenous infusion of Kedrion IVIG 10% at a dose of 200 to 800 milligram per kilogram (mg/kg) body weight every 21 or 28 days for period of 48 weeks.
  Interventions: Biological: Kedrion IVIG 10%

INTERVENTIONS:
Biological: Kedrion IVIG 10% — Kedrion intravenous immunoglobulin (IVIg) 10%

SUMMARY:
The purpose of this study is to assess efficacy, safety and pharmacokinetics of Kedrion Immunoglobulin 10% (KIg10) in pediatric patients with Primary Immunodeficiency Disease (PID).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent obtained from the patient and his/her parent(s) or legally acceptable representative indicating that they understand the purpose of and procedures required for the study and are willing to participate in it.
2. Confirmed clinical diagnosis of a PID as defined by 2017 International Union of Immunological Societies (IUIS) Phenotypic Classification for Primary Immunodeficiencies (Bousfiha A, 2018 - and subsequent revisions) and The European Society for Immunodeficiencies (ESID) Registry Working Definitions for the Clinical Diagnosis of Inborn Errors of Immunity (Seidel MG et al., 2019 - and subsequent revisions) and requiring treatment with IVIg. Documented agammaglobulinemia (defined as the total absence of one or more classes of antibodies) or hypogammaglobulinemia (defined as low levels of one or more classes [i.e., at least 2 standard deviations under the mean level per age]).

   (NOTE: IVIg treatment is generally requested in the absence of IgG independently from whether other antibodies are absent).
3. Male or female, age from 2 up to < 16 years, at the time of screening.
4. Received 200 to 800 mg/kg of a commercially available IVIg therapy in the range of 21- or 28-day intervals (±3 or ±4 days, respectively) for at least 3 infusions prior to screening.

   (NOTE: Other IVIgs will be prohibited after ICF signature and until study end, week 51/52).
5. At least 2 documented IgG trough levels while receiving an IVIg, of ≥ 6 g/L obtained at 2 infusions within 12 months (1 must be within 6 months) prior to ICF signature.
6. Patient and his/her parent(s)/legal guardian(s) are willing to comply with all requirements of the protocol.
7. Females of child-bearing potential with a negative pregnancy test (serum or urine) and who agree to employ adequate birth control measures during the study, such as:

   1. sexual abstinence, to be evaluated in relation to the preferred and usual lifestyle of the subject;
   2. male or female condom with or without spermicide;
   3. cap, diaphragm or sponge with spermicide;
   4. progestogen-only oral hormonal contraception, if already used in the past on medical prescription.

   Adequate birth control measures should be maintained throughout the study under parental control.
8. Authorization to access personal health information.
9. Patients previously participating in a clinical trial with another experimental IVIg may be enrolled if they have received stable commercially available IVIg therapy for at least 3 infusions (21 or 28 days) prior to screening.
10. Patients currently on treatment with any subcutaneous immunoglobulin (SCIG) can be enrolled if they are switched to stable commercially available IVIg therapy for at least 3 infusions (21 or 28 days) prior to screening.
11. Males or females with a body weight greater than or equal to 15 kg (≥ 15 kg).

Exclusion Criteria:

1. Newly diagnosed PID and naïve to IgG replacement therapy.
2. Dysgammaglobulinemia (defined as a deficiency in one or more classes of antibodies, but not severe enough to require substitutive therapy) or isolated IgG subclass deficiency, or profound primary T cell deficiency (defined as the absence or severe reduction of T lymphocytes [CD3+ < 300 cell/mm3] and an absent or particularly low proliferative response [10% of the lower normal range] to phytohaemagglutinin P [PHA]).
3. History of severe or serious reactions or hypersensitivity to IVIg or other injectable forms of IgG.
4. History of thrombotic events including deep vein thrombosis, cerebrovascular accident, pulmonary embolism, transient ischemic attacks, or myocardial infarction, as defined by at least 1 event in patient's lifetime.
5. IgA deficiency with documented antibodies to IgA.
6. Received blood products that have not undergone viral inactivation measures within 12 months prior to ICF signature.
7. Significant protein losing enteropathy, nephrotic syndrome, or lymphangiectasia.
8. An acute infection as documented by culture or diagnostic imaging and/or a body temperature ≥38.5 °C (≥101.3 °F) within 7 days prior to screening.
9. Acquired immunodeficiency syndrome (AIDS) and/or hepatitis B/C active disease at ICF signature.
10. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times of the upper limit of normal for the laboratory designated for the study.
11. Using an implanted venous access device.
12. Moderate or severe anemia, defined according to patient's age as shown in the following table (World Health Organization, 2011) or persistent severe neutropenia (≤ 500 neutrophils per mm3) or persistent lymphopenia of less than 500 cells per microliter.
13. A severe chronic condition such as renal failure [defined as abnormalities in kidney structure or function that are present for more than 3 months and have health implications. The disease is classified on the basis of cause and category of glomerular filtration rate (GFR) (G1 to G5) and albuminuria (A1 to A3) (KIDIGO, 2017). See the following table], congestive heart failure (New York Heart Association III/IV), cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g., atrial fibrillation), unstable or advanced ischemic heart disease, hyperviscosity, or any other condition that the Investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial.
14. History of a malignant disease other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin within 24 months prior to ICF signature.
15. History of pharmacoresistant epilepsy or multiple episodes of migraine (defined as at least 1 episode within 6 months of ICF signature) not controlled by medication.
16. Patient must not be receiving the following medication from at least 30 days prior to ICF signature:

    1. Steroids, inhaled, oral or parenteral, at a daily dosage of ≥ 0.15 mg/kg/day of prednisone or equivalent).
    2. Other immunosuppressive drugs (including monoclonal antibodies) or chemotherapy.
17. Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Women who become pregnant during the study will be withdrawn from the study.
18. Participated in another clinical study within 30 days prior to ICF signature.
19. Active drug or alcohol abuse or history of drug or alcohol abuse within the 6 months before screening.
20. Direct relative of an employee of the CRO, the study site, or Kedrion.
21. Previously treated under this protocol.
22. Unable to provide informed consent.
23. Patients with any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives or the patient's participation in this trial.
24. Patients with Hypersensitivity to the active substance or to any of the excipients.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Acute Serious Bacterial Infections | From Baseline (Day 1) up to week 51/52
  Incidence rate (i.e., the mean number of acute serious bacterial infections per patientyear) of acute serious bacterial infections (bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis) according to pre-specified criteria).

SECONDARY OUTCOMES:
Serum Immunoglobulin G (IgG) trough levels | Before each infusion of KIg10 and at the study termination visit (Week 51/52)
Immunoglobulin G (IgG) subclasses levels (IgG1, IgG2, IgG3, IgG4) | Before infusions 1, 5, 9 and 13 for the 28-day infusion schedule, and before infusions 1, 7, 11 and 17 for the 21-day infusion schedule
Frequency of patients with total Immunoglobulin G (IgG) below 6 g/L | Day 1 up to week 51/52
Anti-tetanus toxoid antibody level | Before infusions 1, 5, 9 and 13 for the 28-day infusion schedule and before infusions 1, 7, 11 and 17 for the 21-day infusion schedule
  The quantitative evaluation will be reported
Anti-pneumococcal capsular polysaccharide antibody level | Before infusions 1, 5, 9 and 13 for the 28-day infusion schedule and before infusions 1, 7, 11 and 17 for the 21-day infusion schedule
  The quantitative evaluation will be reported
Anti-measles antibody level | Before infusions 1, 5, 9 and 13 for the 28-day infusion schedule and before infusions 1, 7, 11 and 17 for the 21-day infusion schedule
  The quantitative evaluation will be reported
Anti-Haemophilus influenza type b antibody level | Before infusions 1, 5, 9 and 13 for the 28-day infusion schedule and before infusions 1, 7, 11 and 17 for the 21-day infusion schedule
  The quantitative evaluation will be reported
Incidence rate (i.e., the mean number per patient-year) of any infection other than acute serious bacterial infections | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Duration of any infection other than acute serious bacterial infections | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Incidence rate (i.e. the mean number per patient-year) of fever episodes | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Duration of fever episodes | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Overall hospitalization days | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Days of hospitalizations due to infection | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Incidence rate (i.e. the mean number per patient-year) of patient on antibiotics for the treatment of any kind of infection | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Duration of patients on antibiotics for the treatment of any kind of infection | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Days of missed work/school/other major activities due to infections | From day 1 to week 51/52
  Information reported by participant/participant's parent(s)/legal guardian(s) in the Patient Diary, provided starting from the first infusion.
Pediatric Quality of Life Inventory (Pedsql) Score | At baseline, week 24, and study termination visit
  The PedsQL™ Measurement Model is a modular approach to measuring health-related QoL in healthy children and adolescents and those with acute and chronic health conditions. The 23-item PedsQL™ Generic Core Scales were designed to measure the core dimension of health as delineated by the World Health Organization, as well as role (school) functioning.
  The total scale score (23 items) consists of Physical health summary score (8 items) and Psychosocial health summary score (15 items). Physical health summary includes Physical Functioning (8 items) and Psychosocial health summary score includes Emotional Functioning (5 items), Social Functioning (5 items) and School Functioning (5 items). The overall range for PedsQL scores is 0 to 100, with a higher score indicating better quality of life.
Number of Adverse Events (%) and proportion of patients experiencing at least one Adverse Event (AE) | From Baseline (Day 1) up to Week 51/52
Number of Serisous AEs (%) and proportion of patients experiencing at least one Serious Adverse Event (SAE) | From Baseline (Day 1) up to Week 51/52
Number of related infusion AEs (%) occurring during infusion or within 1, 24, and 72 hours after the end of infusion, and proportion of patients experiencing at least one related infusion AE. at least 1 of such related infusion AE. | From Baseline (Day 1) up to Week 51/52
The proportion and number of KIg10 infusions for which the infusion rate is decreased due to Adverse Events. | From Baseline (Day 1) up to Week 51/52
Number and proportion of infusions with one or more infusion (temporally-associated) Adverse Event. | From Baseline (Day 1) up to Week 51/52
Number of Participants with Changes from Baseline Values in Vital Signs, Physical Examinations, Safety Laboratory Tests (hematology, serum chemistry and urinalysis). | Up to Week 51/52
  Number of participants with changes from baseline in vital signs (including blood pressure, heart rate and temperature); Physical examination (including evaluation of all body systems, body weight, height and Tanner Staging); Safety Laboratory Tests (including hematology, serum chemistry, and urinalysis) will be reported.
The proportion and number of patients with a positive Coomb's test | Following infusion 7 for the 28-day infusion schedule and infusion 9 for the 21-day infusion schedule
The proportion and number of patients with a positive urine hemosiderin test | Following infusion 7 for the 28-day infusion schedule and infusion 9 for the 21- day infusion schedule
Serum haptoglobin level | Following infusion 7 for the 28-day infusion schedule and infusion 9 for the 21-day infusion schedule.
Serum Total Immunoglobulin G (IgG) levels, IgG Subclasses Levels, and Selected Specific Antibody Levels | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Plasma Concentration - Time Curve Of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Elimination Half-Life (t1/2) of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC(0-T)) of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUC[0-inf]) of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Volume of Distribution of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Maximum Observed Plasma Concentration (Cmax) Of Total IgG | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Time to Reach the Maximum Plasma Concentration (Tmax) of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Elimination Rate Constant of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-Tau) of Total Immunoglobulin G (IgG) | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Plasma Concentration-Time Curve Of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
  The quantitative evaluation of the anti-Tetanus toxoid, anti-pneumococcal capsular polysaccharide, anti-Haemophilus influenza type B and anti-measles antibodies level will be reported
Elimination Half-Life (t1/2) of Specific IgG Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC(0-T)) of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Volume Of Distribution of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Maximum Observed Plasma Concentration (Cmax) of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Time to Reach the Maximum Plasma Concentration (Tmax) of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Elimination Rate Constant of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC[0-inf]) of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)
Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-Tau) of Specific Immunoglobulin G (IgG) Antibodies | Before and after infusion 5 (28-day infusion schedule) or infusion 7 (21-day infusion schedule)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Azzari, Principal Investigator — Azienda Ospedaliero-Universitaria Ospedale Pediatrico Meyer - Italy
Locations (21):
- United States (8):
  - Benioff Children's Hospital - Mission Bay, San Francisco, California
  - IMMUNOe Health and Research Centers, Centennial, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Velocity Clinical Research - MedPharmics - Lafayette, Lafayette, Louisiana
  - Louisiana State University Shreveport, Shreveport, Louisiana
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Asthma and Allergy Center - Toledo, Toledo, Ohio
  - Vital Prospects Clinical Research Institute PC, Tulsa, Oklahoma
- Dél-Pesti Centrumkórház - Országos Hematológiai És Infektológiai Intézet, Budapest, Hungary
- Italy (7):
  - SST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria - Ospedale Pediatrico Meyer, Florence
  - I.R.C.C.S. Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinic, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione Policlinico Tor Vergata, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
- Portugal (2):
  - Centro Hospitalar Lisboa Central - Hospital Dona Estefânia, Lisbon
  - Centro Hospitalar Universitário do Porto - Hospital Santo António, Porto
- Russia (2):
  - Children's City Clinical Hospital No. 9 named after G.N. Speransky, Moscow City Health Department, Moscow
  - Dmitry Rogachev National Medical Research Center for Pediatric Hematology, Oncology and Immunology, Moscow
- Národný ústav detských chorôb (National Institute of Pediatric Diseases), Bratislava, Slovakia